CLINICAL TRIAL: NCT05483283
Title: Empowering Vulnerable and Resilient Latinas to Obtain Breast Cancer Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Yamile Molina, Prinicipal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2022-0378
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Empowerment and navigation and Standard of Care (SOC) (Control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Other): Empowerment and Navigation
  Interventions: Other: Empowerment and Navigation
- Arm 2 (Other): Standard of Care (SOC)
  Interventions: Other: SOC

INTERVENTIONS:
Other: Empowerment and Navigation — Empowerment and Navigation
  Arms: Arm 1
Other: SOC — SOC
  Arms: Arm 2

SUMMARY:
The investigator and study staff will identify, recruit and randomize Latina participants with elevated genetic and Social Determinants of Heath (SDH) risks. Within 1 week of enrollment, all Latina Aim 1 participants in both study arms will engage in three 30-minute, individual, phone-based sessions with the study team across 3 consecutive weeks

DETAILED DESCRIPTION:
The investigator and study staff will identify, recruit and randomize Latina participants with elevated genetic and Social Determinants of Heath (SDH) risks. Within 1 week of enrollment, all Latina Aim 1 participants in both study arms will engage in three 30-minute, individual, phone-based sessions with the study team across 3 consecutive weeks. Sessions will be based on landline or cellphone calls. Within 1 week after each session, all Latina Aim 1 participants will receive copies of the multi-media materials (e.g., personalized plans) by text message or mail, depending on participants' preferences

Control Sessions will be as follows:

Session 1 Learning about Breast Cancer (BC) care uptake Targets the effects of Social Determinants of Heath (SDH) and genetic risk factors on Non-Latino White (NLW) Latino BC disparities Study staff will give personnel testimonials, empirical data and individual action plans behavior change and BC care uptake Session 2 Learning about Diet to promote BC prevention per the American Cancer Society (ACS) BC screening and prevention guidelines Session 3 Learning about Physical Activity to promote BC prevention

Empowerment and Navigation Sessions will be as follows:

Session 1 Learning about Breast Cancer (BC) care uptake Targets the effects of SDH and genetic risk factors on NLW/Latino BC disparities ACS BC screening and prevention guidelines Identify and address SDH and genetic risk factors Study staff will give personnel testimonials, empirical data and individual action plans for behavior change Session 2 Teaching about BC Targets the importance of sharing BC information and personal barriers & preferred solutions to sharing BC information Study staff will give personnel testimonials and individual action plans for sharing information and role playing activities Session 3 Teaching about BC Targets opportunities & skills in sharing BC information participants will give testimonials and relay empirical data. There will be a group discussion and plans for sharing information

There will be a post intervention BC survey call and an end of study BC survey call

Bicultural, bilingual study staff will engage participants in a 5-10 minute call/text every month to "check in" until the end of the study

ELIGIBILITY:
Inclusion Criteria:

Aim 1

1. female biological sex
2. identification as Latina
3. one genetic risk factor (i.e., personal history of breast cancer or family history of breast or ovarian cancer)
4. one SDH risk factor, based on the American Cancer Society's definitions (e.g., perceived financial struggles; transportation difficulties; exposure to violence; housing challenges; social isolation/challenges)
5. 30+ years old, based on American Cancer Society (ACS) screening guidelines for high risk populations
6. No receipt of cancer genetic counseling AND no receipt of genetic testing

Aim 2

1. female biological sex
2. referral from Latina Aim 1 participants
3. eligibility to obtain BC screenings, based on ACS guidelines (e.g., optional annual
4. screenings at 40-44 years old, recommended annual screenings at 45-54 years old, every other year screening at 55 and older)
5. self-report not attending Session #3 (as this will not be recorded by the staff)

Aim 3

1. participant from Aim 1 or
2. participant from Aim 2

Exclusion Criteria:

Aim 1 and Aim 2 Not meeting at least one of the inclusion criteria

Aim 3

1. Not a participant from Aim 1 or
2. Not a participant from Aim 2

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Empower and navigation versus SOC | 4 years
  Number of participants that undergo risk-based BC screening per ACS guidelines versus the control group
Empower and navigation versus SOC | 4 years
  Number of participants that undergo recommended genetic services versus the control group

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Chicago, Illinois, United States